CLINICAL TRIAL: NCT03332446
Title: Influence of Cooling on the Effect of Strength Training
Acronym: IceAge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Anne Krieg M.D., Medical Doctor and Researcher, Universität des Saarlandes
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2512BI1901
Record Dates: First submitted 2016-03-29; First posted 2017-11-06 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Strength Training Effects
Keywords: cold water immersion, strength training, training effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cooling (Experimental): strength training and cold water immersion
  Interventions: Other: cold water immersion
- control (No Intervention): strength training and no cold water immersion

INTERVENTIONS:
Other: cold water immersion — 10 min at 12-15°C
  Arms: cooling

SUMMARY:
The aim of this study is to investigate if regular cold water immersion after strength training has a negative influence on the desired training-induced performance enhancement.

DETAILED DESCRIPTION:
Recovery strategies represent a not sufficiently investigated chance in elite training control to optimize the complete training process. Coaches and athletes are confronted with numerous potentially effective recovery methods, e.g. cooling, warming, active recovery, compression, massage or power naps. However, the effectivity of these methods has rarely been investigated under controlled scientific conditions. Based on the state of the art,so far hardly any definite practical conclusions regarding effective recovery methods can be drawn, especially regarding sport-specific strategies and settings. Currently, cold water immersion is a particularly popular recovery strategy. However, there are hints that repeated cooling interventions after training can impair the training effect. This could potentially be caused by a faster reconstitution of homeostasis due to cooling. For fast recovery of performance, this effect would be desirable, but at the same time these homeostatic disturbances are the basis of signal processes leading to training adaptations.

The aim of this study is to investigate if regular cold water immersion after strength training has a negative influence on the desired training-induced performance enhancement.

ELIGIBILITY:
Inclusion Criteria:

* healthy, 18-40 years, strength training experience, 8 weeks no leg strength training

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-08; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
1 Repetition Maximum | 8 weeks
  Maximum weight in kg that can be successfully moved in a leg press

SECONDARY OUTCOMES:
Counter Movement Jump | 8 weeks
  Maximum jump height in cm in a counter movement jump, measured with a force plate
blood parameters | 8 weeks
  CRP, CK, IL-6, IGF-1
muscle biopsy | 8 weeks
  p70S6, PAX7+, NCAM+
muscle thickness | 8 weeks
  upper leg circumference in cm
subjective restfulness of sleep | 2 weeks
  5-point Likert scale on subjective restfulness of sleep (1: very, 5: not at all)
time in bed | 2 weeks
  Questionnaire recording time of going to bed (time in hh:mm), sleep onset latency (duration in min), waking time (time in hh:mm), and time of getting up (time in hh:mm). From these items, the average time in bed per day is calculated, starting at "time of going to bed" and ending at "time of getting up".
sleeping time | 2 weeks
  Questionnaire recording time of going to bed (time in hh:mm), sleep onset latency (duration in min), waking time (time in hh:mm), and time of getting up (time in hh:mm). From these items, the average sleeping time per day is calculated, starting at "time of going to bed + sleep onset latency" and ending at "waking time".
questionnaire on recovery and stress | 2 weeks
  Short Recovery and Stress Scale for Sport (SRSS): assessing recovery (physical performance capability, mental performance capability, emotional balance, overall recovery) and stress (muscular stress, lack of activation, negative emotional state, overall stress), each item is rated on a 7-point rating scale (0: does not apply at all, 6: fully applies). For evaluation, two outcome values ("recovery" and "stress") are calculated as the sum of the corresponding subvalues, i.e. each outcome value is on a 25-point scale (0: does not apply at all, 24: fully applies).

CONTACTS AND LOCATIONS:
Overall Officials: Tim Meyer, Prof., Principal Investigator — Universität des Saarlandes
Locations (1):
- Saarland University, Saarbrücken, Saarland, Germany

IPD SHARING:
Plan to Share IPD: Undecided